CLINICAL TRIAL: NCT04218903
Title: Comparison of Different Weekly Frequencies of Combined Training on Ambulatory Blood Pressure and Other Cardiovascular Risk Factors in Individuals With Hypertension: a Randomized Clinical Trial
Brief Title: Resistance Plus Aerobic Training Using Different Weekly Frequencies And Hypertension
Acronym: RADAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19816719900005327
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Cardiovascular Risk Factor; Cardiovascular Diseases
Keywords: Aging; Ambulatory Blood Pressure Monitoring; Concurrent Training; Dose-response
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — CD5L protein, human

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Training 4 times per week (CT4) (Experimental): The CT4 group will perform four sessions per week of combined exercise program. This intervention will last 12 weeks.
  Interventions: Behavioral: Combined training performed four times per week (CT4)
- Combined Training 2 times per week (CT2) (Active Comparator): The CT2 group will perform two sessions per week of combined exercise program. This intervention will last 12 weeks.
  Interventions: Behavioral: Combined training performed two times per week (CT2)

INTERVENTIONS:
Behavioral: Combined training performed four times per week (CT4) — CT4 will perform four combined training sessions per week throughout 12 weeks. Each session will be composed 10-15 minutes of resistance exercise (1-4 sets of 10-15 repetitions, using an intensity corresponding to 50-70%1RM in 3 exercises) followed by 20-25 minutes of aerobic exercise (walking or running at an intensity corresponding to 60-70% of VO2peak).
  Arms: Combined Training 4 times per week (CT4)
Behavioral: Combined training performed two times per week (CT2) — CT2 will perform two combined training sessions per week throughout 12 weeks. Each session will be composed 20-30 minutes of resistance exercise (1-4 sets of 10-15 repetitions, using an intensity corresponding to 50-70%1RM in 6 exercises) followed by 40-50 minutes of aerobic exercise (walking or running at an intensity corresponding to 60-70% of VO2peak).
  Arms: Combined Training 2 times per week (CT2)

SUMMARY:
Combined training is a cornerstone intervention to improve functionality and to reduce blood pressure in older adults with hypertension. Acute blood pressure lowering after exercise seems to predict the extent of blood pressure reduction after chronic training interventions. Based on that, the same weekly amount of exercise performed more frequently could be more beneficial to blood pressure management. The aim of the present study is to evaluate the effects of a combined exercise program performed four versus two times per week on 24-h ambulatory blood pressure and other cardiovascular risk factors in older individuals with hypertension.

DETAILED DESCRIPTION:
Chronic blood pressure reduction due regular exercise seems to result from the sum of the acute decreases that follows each exercise bout (i.e., post-exercise hypotension), a physiological effect associated with chronic blood pressure reduction that may predict the extent of blood pressure lowering after chronic training interventions. Based on this, the same weekly amount of exercise performed more frequently, splitting the total overload into multiple sessions, could be more beneficial for blood pressure control. Although physical exercise guidelines suggest a total weekly volume in minutes (i.e., 150 minutes per week), it's unclear if the same amount of exercise performed in different weekly frequencies could induce different blood pressure responses.

The aim of the present study is to evaluate the effects of a combined exercise program performed four versus two times per week on 24-h ambulatory blood pressure and other cardiovascular risk factors in middle-aged and older individuals with hypertension. The main outcome is the change from baseline to 12 weeks of follow-up in 24-h, daytime, nighttime systolic and diastolic ambulatory blood pressure.

Secondary outcomes are the difference between mean change in office blood pressure, cardiorespiratory fitness, muscular strength and quality of life. We anticipate that at 12 weeks, combined exercise program, performed four or two times per week with equalized weekly volume/overload, will improve all outcomes in comparison to the baseline values and these improvements in blood pressure will be more pronounced in four times per week group when compared with two times per week group.

This study will be a randomized, parallel group, two-arm, superiority trial. Ninety-eight participants aged 50-80 years with a previous physician diagnosis of hypertension will be randomized to perform two or four sessions per week of combined training using the same total weekly overload. Primary outcomes will be 24-h ambulatory blood pressure; secondary outcomes will be office blood pressure, physical fitness and quality of life. The outcomes will be assessed at baseline and at the end of 12 weeks period.

ELIGIBILITY:
Inclusion Criteria:

Office blood pressure between 130-179 and 80-110 mmHg for systolic and diastolic blood pressure, respectively or taking at least one antihypertensive medication

Not engaged in structured exercise programs (3 or more times per week) in the last 3 months before the study

Exclusion Criteria:

Physical and muscular injuries that limit to accomplishment of the different training proposed in the study

Underlying cardiovascular disease in the last 24 months such as acute myocardial infarction, angina, stroke or heart failure

Health conditions that limit physical exercise perform, such as lung disease, valvar heart disease, renal failure

Diseases that reduce life expectancy

BMI > 39.9 kg/m²

Diabetic proliferative retinopathy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure | Change from baseline 24-hour systolic blood pressure at 12 weeks
  24h ambulatory blood pressure measured through automatic oscillometric device

SECONDARY OUTCOMES:
Systolic blood pressure | Change from baseline office blood pressure at 12 weeks
  Systolic blood pressure in mmHg measured using automatic oscillometric device
Diastolic blood pressure | Change from baseline office blood pressure at 12 weeks
  Diastolic blood pressure in mmHg measured using automatic oscillometric device
Cardiorespiratory fitness | Change from baseline VO2peak at 12 weeks
  Oxygen consumption at peak (VO2peak) was assessed by maximal cardiopulmonary exercise testing
Upper limbs muscle strength | Change from baseline handgrip test at 12 weeks
  Performs palmar grip with the greatest possible force
Lower limbs muscle strength | Change from baseline sitting-rising test at 12 weeks
  Sitting-rising test in a chair (maximum number of repetitions in 30 seconds and time to 5-repetions)
Quality of life profile | Change from baseline quality of life score at 12 weeks
  World Health Organization Quality of Life questionnaire (WHOQOL-BREF) contains 26 questions using a likert scale (scores range 1 to 5) and has been stratified in 4 domains (physical health, psychological, social relationships and environment). Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ferrari, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided